CLINICAL TRIAL: NCT02422966
Title: Efficacy and Safety of Paracetamol in Comparison to Ibuprofen for Patent Ductus Arteriosus Treatment in Preterm Infants: A Randomized, Open Label, Comparator-controlled, Prospective Study
Brief Title: Paracetamol in Patent Ductus Arteriosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 044CF13273
Record Dates: First submitted 2015-04-09; First posted 2015-04-22 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Ductus Arteriosus, Patent
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracetamol (Experimental): Paracetamol intravenous solution 15 mg/kg (corresponding to 1.5 ml/kg) per dose every 6 hours for 3 days, for a total amount of 12 doses.
  Interventions: Drug: Paracetamol
- Ibuprofen (Active Comparator): Ibuprofen intravenous solution at an initial dose of 10 mg/kg, followed by 5 mg/kg at 24 and 5 mg/kg at 48 h.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Paracetamol
  Other Names: Acetaminophen
  Arms: Paracetamol
Drug: Ibuprofen
  Arms: Ibuprofen

SUMMARY:
The purpose of the study is to assess the efficacy and safety of paracetamol in comparison to ibuprofen in the treatment of patent ductus arteriosus (PDA) in preterm infants.

DETAILED DESCRIPTION:
Although patency of the ductus arteriosus is essential for fetal circulation, the postnatal ductal closure is critical for postnatal circulatory adaptation. In premature infants the circulating prostaglandin levels are higher than at term, and respiratory difficulties may lead to a state of hypoxia, which contribute to the failure of the ductus closure. Recently, an incidental finding in one preterm infant led to look at paracetamol, one of the most common drugs available, as an alternative therapeutic approach to ductal closure. If paracetamol is proven to be effective, it could become the treatment of choice for the management of PDA, mainly due to its more favorable safety profile.

Although the recent results available in the literature demonstrates an highly success rate in ductal closure with paracetamol, all case studies are not powered to show efficacy of paracetamol for PDA closure. Further prospective randomized-controlled trials are needed to evaluate the efficacy of paracetamol versus ibuprofen for the closure of PDA.

If paracetamol is indeed proven to be effective, it could become the treatment of choice for the management of PDA, mainly due to its more favorable side effect profile. In order to test this hypothesis, a randomized, open label, parallel groups, comparator controlled, multicentre, prospective study is proposed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female preterm infants with no limitation of race.
2. Gestational age 25(+0) - 31(+6) weeks.
3. Age 24-72 hours.
4. Echocardiographic evidence of hemodynamically significant patent ductus arteriosus at the first 24-72 hours of life.

   The diagnosis of hemodynamically significant PDA requiring treatment will be made by echocardiographic demonstration of a ductal left-to-right shunt, with a left atrium-to-aortic root ratio >1.3 or a ductal size >1.5 mm and excluding the cases in which the closing flow pattern suggests a restrictive PDA.
5. Willingness of the parents/legally authorized representative/child to sign the Consent Informed Form.

Exclusion Criteria:

1. Outborn patients.
2. Major congenital anomalies, including but not limited to congenital heart defects, Down syndrome newborn and/or new born suffering from congenital anomalies diagnosed during the fetal period.
3. Known positive HIV and/or known positive Hepatitis C Virus newborn's mother.
4. Life threatening infection, complicated or not by multiple organ dysfunction and failure syndrome.
5. Fetal hydrops.
6. Pulmonary hypertension diagnosed in the first 24-48 hours of life by means of heart ultrasound when the presence of a right-to-left shunt through the foramen ovale or ductus arteriosus is demonstrated, or when the estimated pulmonary pressure, in terms of the tricuspid regurgitation jet, is greater than two-thirds of the systemic arterial pressure.
7. Grade 3 or 4 intraventricular haemorrhage (IVH).
8. Urine output <1 ml/kg of body weight/h during a 24 h collection period or urine output <0.5 ml/kg of body weight/h in case it is measured at 24 hours of life of newborn.
9. Serum creatinine concentration > 1.5 mg/dl (132 μmol/l).
10. Platelet count < 50,000/mm3.
11. Major bleeding, as revealed by hematuria, or blood in the endotracheal aspirate, gastric aspirate, or stools, or consistent oozing of blood from puncture sites.
12. Severe liver failure, defined as elevated liver enzymes (ALT/Glutamate-Pyruvate Transaminase and Aspartate aminotransferase/GOT) > 2 times the upper boundary of the normal range. For this kind of population the following normal ranges will be considered [Rosenthal, 1997]:

    * ALT/Glutamate-pyruvate transaminase: 6-50 U/L
    * Aspartate aminotransferase/GOT: 35-140 U/L
13. Medical need of administering other Nonsteroidal Antiinflammatory Drug (NSAID) different from ibuprofen.
14. Participation to another trial involving any investigational drug.

Ages: 25 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
success rate in closing PDA using paracetamol in comparison to ibuprofen. | at Visit 3 (day 3).
  assessed echocardiographically.

SECONDARY OUTCOMES:
number of re-openings. | at Follow-up 3 (day 30).
  assessed echocardiographically.
success rate in closing PDA after the second treatment course of ibuprofen as rescue medication. | at Visit 6 (day 6).
  assessed echocardiographically.
success rate of closing PDA after the first day of the first treatment course. | at Visit 1 (day 1).
  assessed echocardiographically.
success rate of closing PDA after the second day of the first treatment course. | at Visit 2 (day 2).
  assessed echocardiographically.
incidence of surgical ligation. | at Follow-up 3 (day 30).
incidence of renal failure, liver failure and gastrointestinal complications (including isolated intestinal perforation). | at Follow-up 3 (day 30).
  assessed by laboratory analysis.
incidence of death, | at Follow-up 3 (day 30).
incidence of death. | at Follow-up 4 (40 weeks post-conception).
incidence of sepsis. | at Follow-up 3 (day 30).
hospital-stay duration in Neonatal Intensive Care Unit. | at Follow-up 4 (40 weeks post-conception).
occurrence of adverse effects. | at Follow-up 3 (day 30).

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Azienda Ospedaliero Universitaria Careggi - Neonatologia e Terapia Intensiva Neonatale, Florence
  - IRCCS "Giannina Gaslini" Genova - Patologia Neonatale e Terapia Intensiva Neonatale, Genova
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico U.O. di Neonatologia e Terapia Intensiva Neonatale, Milan
  - Azienda Ospedaliera Istituti Clinici di Perfezionamento (ICP) - Ospedale dei Bambini "Vittore Buzzi" Milano - Neonatologia, Milan
  - Policlinico Gemelli Roma - UOC Neonatologia, Roma

REFERENCES:
- [Derived] Jasani B, Mitra S, Shah PS. Paracetamol (acetaminophen) for patent ductus arteriosus in preterm or low birth weight infants. Cochrane Database Syst Rev. 2022 Dec 15;12(12):CD010061. doi: 10.1002/14651858.CD010061.pub5. PMID 36519620
- [Derived] Dani C, Lista G, Bianchi S, Mosca F, Schena F, Ramenghi L, Zecca E, Vento G, Poggi C, Leonardi V, Minghetti D, Rosignoli MT, Calisti F, Comandini A, Cattaneo A, Lipone P. Intravenous paracetamol in comparison with ibuprofen for the treatment of patent ductus arteriosus in preterm infants: a randomized controlled trial. Eur J Pediatr. 2021 Mar;180(3):807-816. doi: 10.1007/s00431-020-03780-8. Epub 2020 Sep 4. PMID 32888085
- [Derived] Dani C, Poggi C, Mosca F, Schena F, Lista G, Ramenghi L, Romagnoli C, Salvatori E, Rosignoli MT, Lipone P, Comandini A. Efficacy and safety of intravenous paracetamol in comparison to ibuprofen for the treatment of patent ductus arteriosus in preterm infants: study protocol for a randomized control trial. Trials. 2016 Apr 2;17:182. doi: 10.1186/s13063-016-1294-4. PMID 27038924